CLINICAL TRIAL: NCT01925859
Title: Pharmacokinetics Study to Measure Plasma Concentrations of Dexamethasone Following EryDex (Dexamethasone Sodium Phosphate Encapsulated in Autologous Erythrocytes) Infusion in Healthy Volunteers
Brief Title: EryDex Pharmacokinetics in Healthy Volunteers
Acronym: EryDex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Quince Therapeutics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IED-PK01-2013
Record Dates: First submitted 2013-08-14; First posted 2013-08-20 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: Pharmacokinetic analysis; EryDex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EryDex System (Experimental): erythrocytes encapsulated with dexamethasone sodium phosphate (EryDex System)
  Interventions: Drug: EryDex (dexamethasone sodium phosphate encapsulated erythrocytes)

INTERVENTIONS:
Drug: EryDex (dexamethasone sodium phosphate encapsulated erythrocytes) — erythrocytes encapsulated with dexamethasone sodium phosphate (EryDex System)-corresponding to either 50 mg OR 125mg of experimental study drug
  Other Names: EryDex System (dexamethasone sodium phosphate encapsulated erythrocytes)

SUMMARY:
To compare the pharmacokinetic properties of two different doses of EryDex (dexamethasone sodium phosphate encapsulated in erythrocytes) given as a single infusion in healthy volunteers, based on plasma concentrations of dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-55 years, inclusive.
2. If female, the subject is not pregnant or lactating, and has negative serum pregnancy tests at Screening and Baseline (check-in).
3. If female of childbearing potential*, the subject agrees not to donate ova and to use one of the following methods of contraception from the time of signing the informed consent until 2 months after infusion.

   1. Cap or diaphragm with spermicidal cream or jelly + male condom and spermicide.
   2. Hormonal contraceptives (oral, implant, injection or patch) + male condom and spermicide.
   3. Intrauterine devices + male condom or spermicide.
   4. Vaginal ring + male condom and spermicide.

      * Non-childbearing potential is defined as surgical sterilization (hysterectomy, bilateral oophorectomy, or bilateral tubal ligation), hysterectomy at least 3 months before the start of the study, or postmenopausal (defined as continuous amenorrhea for at least 2 years).
4. If male, the subject agrees to not donate sperm and to use barrier contraception (e.g., condom with spermicidal cream or jelly) from the time of signing the informed consent until 2 months after infusion.
5. Physically and mentally healthy, as confirmed by medical history, physical examination, vital signs, clinical laboratory tests, and ECG.
6. The subject has a body weight of at least 45 kg and a body mass index of ≤ 30.
7. Written informed consent to participate was obtained from the subject.
8. Ability to understand the aims of the trial and comply with the study procedures.

Exclusion Criteria:

* General

  1. Females that are of childbearing potential, pregnant, or are breast-feeding. Women of childbearing potential using two forms of birth control (e.g. barrier and hormonal) will be eligible.
  2. Loss/removal of 500 mL or more of blood within the past 4 weeks.
  3. A disability that may prevent the subject from completing all study requirements.
  4. Noncompliance with the study requirements. Medical History
  5. Current or previous neoplastic disease.
  6. History of any impairment of the immunological system.
  7. History of drug or alcohol abuse (within past 5 years).
  8. A current diagnosis of severe or unstable cardiovascular disease;
  9. Any history or current evidence of a cardiac illness as determined by the investigator;
  10. History or current diagnosis of a psychiatric illness (DSM-IV-TR Axis I diagnosis) or neurodegenerative disorder.
  11. Smoker; currently or at any time in the last 6 months.
  12. Hemoglobinopathy or G6PD deficiency.
  13. History of recurrent or chronic infections, including Staphylococcus or methicillin-resistant Staphylococcus aureus (MRSA).
  14. History of positive tuberculosis skin test (PPD test). Current Medical Status
  15. Have any other significant disease or condition that in the Investigator's opinion would put the subject at risk for participating in the trial.
  16. Vital signs outside the following ranges:

      1. Systolic blood pressure <90 or >140 mmHg
      2. Diastolic blood pressure <50 or >90 mmHg
      3. Pulse <50 or >90 bpm. Patients with pulse rates <50 that are otherwise healthy will be eligible for the trial if approved by the Sponsor.
  17. Any clinically significant ECG abnormality, including a disorder of rate, rhythm, or conduction, or other morphological changes.
  18. Any clinically significant abnormality on standard laboratory examinations (hematology, biochemistry, urinalysis), as determined by the Investigator, in consultation with the Sponsor.
  19. History of hepatitis B and/or C, and/or positive serology results, which indicate the presence of hepatitis B and/or C (Hepatitis B surface antigen and/or antibody to Hepatitis C).
  20. Positive results from the HIV serology.
  21. Positive results of the drug and alcohol tests at screening and/or check-in at the unit. Alcohol intake should be limited to 2 drinks per day during the 2 weeks prior to dosing; alcohol consumption will be prohibited from the time o
  22. Clinically significant abnormal serum cortisol levels (below normal range or >1.5x ULN) at screening.

      Prior/Concomitant Medication
  23. Any previous steroid consumption within 4 weeks before Baseline.
  24. Chronic condition or prior allergic reaction representing a contraindication to the use of steroid drugs.
  25. Have participated in any other trial with an investigational drug and received a dose within 30 days or 10 half-lives (whichever is greater) from the start of the Screening Period.
  26. Requirement for any prescription or over-the-counter (OTC) medication, other than hormonal birth control or occasional use of acetaminophen, that cannot be discontinued during screening, at least one week before Baseline, and throughout the 42-day study period.

      f admittance on Day -1 through to the final safety evaluations on Day 42.
  27. A drug or treatment known to cause major organ system toxicity during the past year.
  28. Caffeine-containing products in excess of the equivalent of 2 cups of coffee per day during the 2 weeks prior to dosing and through to the final safety evaluations on Day 42.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic comparison of two different doses of EryDex in two independent groups | 42 days after infusion
  • To compare the pharmacokinetic (PK) properties of 2 different doses of EryDex (dexamethasone sodium phosphate encapsulated in erythrocytes) given as a single infusion in healthy volunteers, based on plasma concentrations of dexamethasone.

SECONDARY OUTCOMES:
Evaluation of safety and tolerability of a single infusion of EryDex administered in two different doses in healthy volunteers | 84 days after infusion
  • To evaluate the safety and tolerability of a single infusion of EryDex, administered at 2 different doses in healthy volunteers, based on the following: Treatment-Emergent Adverse Events (TEAEs), Serious AEs (SAEs), laboratory parameters, vital signs, ECGs and physical examination findings.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Ibrahim, MD, Principal Investigator — SNBL Pharmacology Center
Locations (1):
- SNBL Clinical Pharmacology Center, Baltimore, Maryland, United States